CLINICAL TRIAL: NCT03764462
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Characteristics of AD-101 in Healthy Volunteers
Brief Title: Evaluating the Pharmacokinetic Characteristics of AD-101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-101BE
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — AD 101; Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raloxifene 60mg to AD-101 45mg (Experimental): Period 1: Raloxifene 60mg, 1 tab, QD, Per oral / Period 2: AD-101 45mg, 1 tab, QD, Per oral
  Interventions: Drug: AD-101 45mg; Drug: Raloxifene 60mg
- AD-101 45mg to Raloxifene 60mg (Experimental): Period 1: AD-101 45mg, 1 tab, QD, Per oral / Period 2: Raloxifene 60mg, 1 tab, QD, Per oral
  Interventions: Drug: AD-101 45mg; Drug: Raloxifene 60mg

INTERVENTIONS:
Drug: AD-101 45mg — Raloxifene 45mg tablet
  Other Names: AD-101
Drug: Raloxifene 60mg — Raloxifene 60mg tablet

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics of AD-101 in healthy volunteers

DETAILED DESCRIPTION:
This study is to evaluate the pharmacokinetic characteristics and safety of AD-101 compared with administration of raloxifen 60 mg in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult aged 19 and more at the time of screening visit
* Body mass index (BMI) between 17.5 kg/m2 and 30.5 kg/m2 at the time of screening visit
* No evidence of medical symptoms or signs of congenital or no chronic disease within the last 3 years as a result of medical examination

Exclusion Criteria:

* Evidence of clinically significant blood, kidney, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, nerve or allergic disease (except for asymptomatic seasonal allergy untreated at the time of administration)
* History of gastrointestinal disorders (esophageal ataxia or esophageal strictures, Crohn's disease, etc.) or surgery (excluding simple cecal surgery or hernia surgery) that may affect the absorption of drugs
* As a result of laboratory tests, the following figures: ALT or AST> 2 times upper limit of normal range

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | pre-dose to 96 hours
  Cmax of the total ingredient of AD-101
Area under the curve in time plot (AUCt) | pre-dose to 96 hours
  AUCt of the total ingredient of AD-101

SECONDARY OUTCOMES:
Area under the curve in time plot (AUCinf) | pre-dose to 96 hours
  AUCinf of the total ingredient of AD-101
Time to reach Cmax | pre-dose to 96 hours
  Tmax of the total ingredient of AD-101
Effective half-life | pre-dose to 96 hours
  t1/2 of the total ingredient of AD-101
Clearance | pre-dose to 96 hours
  CL/F of the total ingredient of AD-101
Volume of distribution | pre-dose to 96 hours
  Vd/F of the total ingredient of AD-101

OTHER OUTCOMES:
Number of participants with adverse events | From Day 1 until 40 Days
  Incidence rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, M.D., Ph.D, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No